CLINICAL TRIAL: NCT00604175
Title: A Phase II Study to Evaluate the Immunogenicity and Safety of a Quadrivalent Human Papillomavirus Vaccine in HIV-1-Infected Females
Brief Title: Safety of and Immune Response to the Human Papillomavirus (HPV) Vaccine in HIV-Infected Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A5240; 10393 (Registry Identifier: DAIDS ES Registry Number); ACTG A5240
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2015-08

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: HIV; HPV 6; HPV 11; HPV 16; HPV 18; Vaccine
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stratum A (Experimental): Participants with screening CD4 count >350 cells/mm^3 received 0.5mL of quadrivalent HPV vaccine at baseline and Weeks 8 and 24.
  Interventions: Biological: Quadrivalent HPV vaccine
- Stratum B (Experimental): Participants with screening CD4 count >200 to <=350 cells/mm^3 received 0.5mL of quadrivalent HPV vaccine at baseline and Weeks 8 and 24.
  Interventions: Biological: Quadrivalent HPV vaccine
- Stratum C (Experimental): Participants with screening CD4 count <=200 cells/mm^3 received 0.5mL of quadrivalent HPV vaccine at baseline and Weeks 8 and 24.
  Interventions: Biological: Quadrivalent HPV vaccine

INTERVENTIONS:
Biological: Quadrivalent HPV vaccine — Quadrivalent HPV (types 6, 11, 16, 18) recombinant vaccine. All participants received the vaccine via intramuscular injection at baseline, Week 8 and Week 24.
  Other Names: GARDASIL

SUMMARY:
Human papillomavirus (HPV) is the most common sexually transmitted disease in the world. HPV infection can cause genital warts and certain cervical problems, including cervical cancer. HPV infection may be more severe and harder to treat in HIV-infected people. The purpose of this study was to determine whether the quadrivalent HPV vaccine is safe, tolerable, and effective in producing antibodies to HPV in HIV-infected women.

DETAILED DESCRIPTION:
HPV is a DNA virus that affects both men and women. Approximately 90 types of HPV have been identified, 30 of which are sexually transmitted. The most common forms of HPV are types 6, 11, 16, and 18. The quadrivalent HPV vaccine that was tested in this study had been shown in previous studies to be effective in preventing infection with HPV 6, 11, 16, and 18 in healthy young women. According to a report by the Centers for Disease Control and Prevention (CDC), 80% of women will have acquired HPV by the age of 50. HIV infected women have been reported to have a higher prevalence and persistence of HPV infection, as well as an increased risk for abnormal Pap smears and cervical cancer. HPV types 16 and 18 cause the majority of cervical cancers worldwide, and types 6 and 11 are responsible for the majority of cases of genital warts. Vaccinations for preventable infections are particularly important among HIV infected people because people with HIV have compromised immune systems; therefore, any infection is very serious and can potentially be fatal. However, standard vaccination series have not been very successful because a compromised immune system may not produce the desired immune response to a vaccine. The HPV vaccine is designed to protect against infection with HPV types 6, 11, 16, and 18 and has been approved by the FDA for use in women between the ages of 9 and 26. The purpose of this study was to determine whether the quadrivalent HPV vaccine is safe, tolerable, and effective in producing antibodies to HPV in HIV infected females.

The study consisted of single arm evaluations of HPV vaccine immunogenicity and safety in 3 groups based on the study screening CD4 cell count as follows:

* Stratum A: CD4 cell count >350 cells/mm^3
* Stratum B: CD4 cell count >200 to <=350 cells/mm^3
* Stratum C: CD4 cell count <=200 cells/mm^3

In Version 1.0 of the protocol, the target accrual was n=67 participants with screening HIV viral load <=10,000 copies/mL and n=67 participants with HIV viral load >10,000 copies/mL within each CD4 stratum, yielding n=134 in each CD4 stratum. In light of subsequent findings from completed HPV vaccine studies, the sample size was changed to n=94 participants per CD4 stratum in Version 2.0 of the protocol, and stratification by screening HIV viral load was removed. All Stratum A and Stratum B participants were enrolled under protocol Version 1.0.

The study duration was 72 weeks. All participants received HPV vaccine administered by intramuscular injection at baseline, and at Weeks 8 and 24. Following each injection, participants remained at the clinic for 30 minutes of observation for adverse events. A telephone follow-up or a home visit by study staff was performed within 2 days following each injection.

Participants returned to the clinic for visits at Weeks 4, 8, 12, 24, 28, 52, and 72. Most study visits included a physical exam, medication review, blood and urine collection, and answering questions about signs and symptoms since previous visit. Some visits included measurement of HIV viral load and CD4 cell count; collection of endocervical wick, cervical cytobrush and anal swab; and an oral exam. A subset of participants were asked to provide additional blood samples and oral cytobrush specimens.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* CD4 count obtained within 45 days prior to study entry
* Karnofsky performance score >=70 on at least one occasion within 45 days prior to study entry
* The following labs within 45 days prior to study entry:

  * hemoglobin >8.0 g/dL
  * direct bilirubin <2.5 x upper limit of normal (ULN)
  * alanine aminotransferase, ALT (SGPT) <3 xULN
  * aspartate aminotransferase, AST (SGOT) <3 xULN
  * platelet count >=100,000 /mm^3
* Willing to use acceptable forms of contraception for the duration of the study
* Written informed consent from participant or from parent or guardian, if applicable
* If on HAART, then the same regimen for at least 12 weeks prior to study entry with no change within 30 days prior to study entry. (This criterion was removed in Version 2.0 of the protocol.)
* HIV viral load obtained within 45 days prior to study entry (This criterion was removed in Version 2.0 of the protocol.)

Exclusion Criteria:

* Abnormal Pap test with confirmed biopsy results of cervical intraepithelial neoplasia (CIN) II or III or cervical cancer within 180 days prior to study entry
* Vulval intraepithelial neoplasia (VIN) II or III or cancer confirmed by biopsy results within 180 days prior to study entry
* Physician-diagnosed genital warts within 180 days prior to study entry
* Previous cervical dysplasia treatment, including loop electrosurgical excision procedure (LEEP), cervical cryotherapy, cone biopsy, and cervical laser vaporization within 180 days prior to study entry
* Use of any systemic antineoplastic or immunomodulatory treatment, systemic corticosteroids, investigational vaccines, interleukins, interferons, growth factors, or intravenous immunoglobulin (IVIG) within 45 days prior to study entry. Participants who had received standard of care (e.g., hepatitis B, influenza, and tetanus) vaccines were not excluded.
* Known allergy or hypersensitivity to yeast or any components of the vaccine or its formulation
* Current drug or alcohol use or dependence or any other condition that may interfere with study participation
* Serious illness requiring systemic treatment and/or hospitalization within 45 days prior to study entry
* Total hysterectomy. Participants who had undergone partial hysterectomy and had a cervix were not excluded.
* Hemophilia
* Currently on anticoagulation therapy other than acetylsalicylic acid
* Prior vaccination with an HPV vaccine
* Pregnant or breastfeeding

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 319 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erna Milunka Kojic, MD, Study Chair — Department of Immunology/Infectious Disease, The Miriam Hospital, Brown University; Susan Cu-Uvin, MD, Study Chair — Obstetrics-Gynecology and Medicine, The Miriam Hospital, Brown University
Locations (61):
- United States (56):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - Usc La Nichd Crs, Alhambra, California
  - University of California, UC San Diego CRS, La Jolla, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - University of Southern California CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
  - The University of Miami AIDS Clinical Research Unit (ACRU) CRS, Miami, Florida
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Mt. Sinai Hosp. Med. Ctr. - Chicago, Womens & Childrens HIV Program, Chicago, Illinois
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Rush University CRS, Chicago, Illinois
  - Tulane Univ. New Orleans NICHD CRS, New Orleans, Louisiana
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - New Jersey Medical School- Adult Clinical Research Ctr. CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Trillium Health ACTG CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - The Research & Education Group-Portland CRS, Portland, Oregon
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ. Med. Ctr. CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Trinity Health and Wellness Center CRS, Dallas, Texas
  - Texas Children's Hospital CRS, Houston, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia
  - University of Washington AIDS CRS, Seattle, Washington
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro, Brazil
- Puerto Rico (3):
  - Puerto Rico AIDS Clinical Trials Unit CRS, San Juan
  - University of Puerto Rico Pediatric HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan
- Wits Helen Joseph Hospital CRS (Wits HJH CRS), Johannesburg, Gauteng, South Africa

REFERENCES:
- [Background] Cameron JE, Hagensee ME. Human papillomavirus infection and disease in the HIV+ individual. Cancer Treat Res. 2007;133:185-213. doi: 10.1007/978-0-387-46816-7_7. PMID 17672042
- [Background] Chaturvedi AK, Goedert JJ. Human papillomavirus genotypes among women with HIV: implications for research and prevention. AIDS. 2006 Nov 28;20(18):2381-3. doi: 10.1097/01.aids.0000253366.94072.b4. No abstract available. PMID 17117025
- [Background] De Vuyst H, Franceschi S. Human papillomavirus vaccines in HIV-positive men and women. Curr Opin Oncol. 2007 Sep;19(5):470-5. doi: 10.1097/CCO.0b013e3282c8c8fc. PMID 17762573
- [Background] Kojic EM, Cu-Uvin S. Update: human papillomavirus infection remains highly prevalent and persistent among HIV-infected individuals. Curr Opin Oncol. 2007 Sep;19(5):464-9. doi: 10.1097/CCO.0b013e3282c8c84c. PMID 17762572
- [Background] Palefsky J. Human papillomavirus infection in HIV-infected persons. Top HIV Med. 2007 Aug-Sep;15(4):130-3. PMID 17720998
- [Result] Kojic EM, Kang M, Cespedes MS, Umbleja T, Godfrey C, Allen RT, Firnhaber C, Grinsztejn B, Palefsky JM, Webster-Cyriaque JY, Saah A, Aberg JA, Cu-Uvin S. Immunogenicity and safety of the quadrivalent human papillomavirus vaccine in HIV-1-infected women. Clin Infect Dis. 2014 Jul 1;59(1):127-35. doi: 10.1093/cid/ciu238. Epub 2014 Apr 9. PMID 24723284
- [Derived] Kang M, Umbleja T, Ellsworth G, Aberg J, Wilkin T. Effects of Sex, Existing Antibodies, and HIV-1-Related and Other Baseline Factors on Antibody Responses to Quadrivalent HPV Vaccine in Persons With HIV. J Acquir Immune Defic Syndr. 2022 Apr 1;89(4):414-422. doi: 10.1097/QAI.0000000000002891. PMID 34907980
- [Derived] Cespedes MS, Kang M, Kojic EM, Umbleja T, Godfrey C, Webster-Cyriaque JY, Masih R, Firnhaber C, Grinsztejn B, Saah A, Cu-Uvin S, Aberg JA. Anogenital human papillomavirus virus DNA and sustained response to the quadrivalent HPV vaccine in women living with HIV-1. Papillomavirus Res. 2018 Dec;6:15-21. doi: 10.1016/j.pvr.2018.08.002. Epub 2018 Aug 16. PMID 30118852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 319 HIV-infected women 13-45 years of age were recruited in US, South Africa and Brazil between March 2008 and July 2011 for participation in this study.
Pre-assignment Details: Participants were enrolled into 3 strata based on screening CD4 cell count:
  * Stratum A: CD4 cell count >350 cells/mm^3
  * Stratum B: CD4 cell count >200 to <=350 cells/mm^3
  * Stratum C: CD4 cell count <=200 cells/mm^3
Period: Entry Through Week 28
Arm/Group | Stratum A | Stratum B | Stratum C
Started | 130 | 95 | 94
Completed | 120 (Completed 28 weeks of the study (the primary endpoint time point).) | 92 (Completed 28 weeks of the study (the primary endpoint time point).) | 93 (Completed 28 weeks of the study (the primary endpoint time point).)
Not Completed | 10 | 3 | 1
Not completed — Death | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 3 | 0
Not completed — Ineligible | 1 | 0 | 0
Not completed — Did not start intervention | 2 | 0 | 1
Period: Week 29 Through Week 72
Arm/Group | Stratum A | Stratum B | Stratum C
Started | 120 | 92 | 93
Completed | 108 | 85 | 89
Not Completed | 12 | 7 | 4
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 12 | 6 | 2
Not completed — Site closure | 0 | 1 | 0
Not completed — Non-adherence to study requirements | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants, except 4: one was found to be ineligible after enrollment (Stratum A) and 3 failed to start intervention (2 in Stratum A, 1 in Stratum C).
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum A | Stratum B | Stratum C | Total
Number analyzed (Participants) | 127 | 95 | 93 | 315
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [29 to 40] | 38 [33 to 42] | 36 [31 to 40] | 36 [30 to 41]
Age, Customized [Number; unit: Participants]
  13 - 17 years | 0 | 0 | 1 | 1
  18 - 24 years | 10 | 3 | 7 | 20
  25 - 29 years | 24 | 11 | 12 | 47
  30 - 34 years | 26 | 14 | 20 | 60
  35 - 39 years | 31 | 26 | 24 | 81
  40 - 45 years | 36 | 41 | 29 | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 95 | 93 | 315
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Race/ethnicity, self-reported (NIH categories).
  Participants
    White, Non-Hispanic | 19 | 9 | 8 | 36
    Black, Non-Hispanic | 67 | 59 | 51 | 177
    Hispanic (Regardless of Race) | 39 | 25 | 32 | 96
    Asian, Pacific Islander | 2 | 0 | 1 | 3
    Unknown | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: Participants]
  United States | 113 | 80 | 69 | 262
  Brazil | 11 | 6 | 11 | 28
  South Africa | 3 | 9 | 13 | 25
HIV Antiretroviral Therapy (ART) Status [Number; unit: Participants]
  On ART | 58 | 71 | 80 | 209
  Not on ART | 69 | 24 | 13 | 106
CD4 Cell Count [Median (Inter-Quartile Range); unit: Cells/mm^3] | 519 [418 to 664] | 287 [246 to 344] | 154 [86 to 188] | 310 [197 to 498]
Nadir CD4 Cell Count [Median (Inter-Quartile Range); unit: Cells/mm^3] | 368 [234 to 482] | 176 [64 to 261] | 41 [20 to 108] | 179 [47 to 314]
HIV Viral Load [Number; unit: Participants] — A blood sample was drawn for HIV viral load testing by local laboratories. The assays used were Roche Amplicor Monitor HIV RT PCR, Roche UltraSensitive HIV RT PCR, bDNA (Versant HIV-1 RNA 3.0, 3rd), Roche COBAS AmpliPrep/Taqman HIV and Abbott RealTime HIV-1.
  Participants
    <=10,000 copies/mL | 71 | 69 | 61 | 201
    >10,000 copies/mL | 56 | 25 | 32 | 113
    Unknown | 0 | 1 | 0 | 1
Human Papillomavirus Type 6 (HPV6) Serostatus [Number; unit: Participants] — HPV serotyping was performed centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. Seronegative status was defined as HPV6 antibody titers <20 mMU/mL and seropositive as HPV6 antibody titers >=20 mMU/mL.
  Participants
    Seronegative | 66 | 60 | 56 | 182
    Seropositive | 54 | 35 | 37 | 126
    Unknown | 7 | 0 | 0 | 7
Human Papillomavirus Type 11 (HPV11) Serostatus [Number; unit: Participants] — HPV serotyping was performed centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. Seronegative status was defined as HPV11 antibody titers <16 mMU/mL and seropositive as HPV11 antibody titers >=16 mMU/mL.
  Participants
    Seronegative | 99 | 72 | 74 | 245
    Seropositive | 22 | 23 | 19 | 64
    Unknown | 6 | 0 | 0 | 6
Human Papillomavirus Type 16 (HPV16) Serostatus [Number; unit: Participants] — HPV serotyping was performed centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. Seronegative status was defined as HPV16 antibody titers <20 mMU/mL and seropositive as HPV16 antibody titers >=20 mMU/mL.
  Participants
    Seronegative | 77 | 65 | 67 | 209
    Seropositive | 44 | 30 | 26 | 100
    Unknown | 6 | 0 | 0 | 6
Human Papillomavirus Type 18 (HPV18) Serostatus [Number; unit: Participants] — HPV serotyping was performed centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. Seronegative status was defined as HPV18 antibody titers <24 mMU/mL and seropositive as HPV18 antibody titers >=24 mMU/mL.
  Participants
    Seronegative | 92 | 83 | 73 | 248
    Seropositive | 29 | 12 | 20 | 61
    Unknown | 6 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HPV6 Antibody Development From Seronegative Status at Baseline to Seropositive Status a Month After Completion of HPV Vaccination Series
Description: Percentage of participants with HPV6 antibody development from seronegative status (HPV6 antibody titers <20 mMU/mL) at baseline to seropositive (HPV6 antibody titers >=20 mMU/mL) status a month after the completion of HPV vaccination series. HPV serotyping was performed centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum.
Time Frame: Week 28
Population: Per-protocol analysis including all participants seronegative to HPV6 at baseline who completed the vaccination series per protocol and had HPV6 titer available at Week 28.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 54 | 50 | 45
Percentage of participants | 96.3 [87.3 to 99.5] | 100.0 [92.9 to 100.0] | 84.4 [70.5 to 93.5]

2. Primary Outcome: Percentage of Participants With HPV11 Antibody Development From Seronegative Status at Baseline to Seropositive Status a Month After Completion of HPV Vaccination Series
Description: Percentage of participants with HPV11 antibody development from seronegative status (HPV11 antibody titers <16 mMU/mL) at baseline to seropositive (HPV11 antibody titers >=16 mMU/mL) status a month after the completion of HPV vaccination series. HPV serotyping was performed centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum.
Time Frame: Week 28
Population: Per-protocol analysis including all participants seronegative to HPV11 at baseline who completed the vaccination series per protocol and had HPV11 titer available at Week 28.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 86 | 59 | 62
Percentage of participants | 97.7 [91.9 to 99.7] | 98.3 [90.9 to 100.0] | 91.9 [82.2 to 97.3]

3. Primary Outcome: Percentage of Participants With HPV16 Antibody Development From Seronegative Status at Baseline to Seropositive Status a Month After Completion of HPV Vaccination Series
Description: Percentage of participants with HPV16 antibody development from seronegative status (HPV16 antibody titers <20 mMU/mL) at baseline to seropositive (HPV16 antibody titers >=20 mMU/mL) status a month after the completion of HPV vaccination series. HPV serotyping was performed centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum.
Time Frame: Week 28
Population: Per-protocol analysis including all participants seronegative to HPV16 at baseline who completed the vaccination series per protocol and had HPV16 titer available at Week 28.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 67 | 56 | 56
Percentage of participants | 98.5 [92.0 to 100.0] | 98.2 [90.4 to 100.0] | 92.9 [82.7 to 98.0]

4. Primary Outcome: Percentage of Participants With HPV18 Antibody Development From the Seronegative Status at Baseline to Seropositive Status a Month After Completion of HPV Vaccination Series
Description: Percentage of participants with HPV18 antibody development from seronegative status (HPV18 antibody titers <24 mMU/mL) at baseline to seropositive (HPV18 antibody titers >=24 mMU/mL) status a month after the completion of HPV vaccination series. HPV serotyping was performed centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum.
Time Frame: Week 28
Population: Per-protocol analysis including all participants seronegative to HPV18 at baseline who completed the vaccination series per protocol and had HPV18 titer available at Week 28.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 78 | 71 | 61
Percentage of participants | 91.0 [82.4 to 96.3] | 84.5 [74.0 to 92.0] | 75.4 [62.7 to 85.5]

5. Secondary Outcome: HPV6 Antibody Titers Among Those Seronegative for HPV6 at Baseline
Description: HPV antibody titers to type 6 were measured centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. The results below the lower limit of detection (LLD) were assigned the values of half the LLD (7 mMU/mL, and after assay change in December 2012, 11 mMU/mL for HPV6). Geometric mean HPV6 titers with 95% CIs were calculated among the subset of participants who were seronegative for HPV6 (<20 mMU/mL) at baseline.
Time Frame: Weeks 28, 72
Population: All eligible participants who received at least one vaccine and were seronegative for HPV6 (HPV6-) at baseline (the number of participants analyzed) and had HPV6 titer available at the respective follow-up week. Strata A; B; C. Week 28: n=60; 58; 52. Week 72: n=55; 53; 53.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- Stratum A/Baseline HPV6-: Participants with screening CD4+ count >350 cells/mm^3 (Stratum A) who were seronegative for HPV6 at baseline.
- Stratum B/Baseline HPV6-: Participants with screening CD4+ count >200 to <=350 cells/mm^3 (Stratum B) who were seronegative for HPV6 at baseline.
- Stratum C/Baseline HPV6-: Participants with screening CD4+ count<=200 cells/mm^3 (Stratum C) who were seronegative for HPV6 at baseline.
Arm/Group | Stratum A/Baseline HPV6- | Stratum B/Baseline HPV6- | Stratum C/Baseline HPV6-
Number analyzed (Participants) | 66 | 60 | 56
mMU/mL
  HPV6 titers at Week 28 (n=60; 58; 52) | 462.3 [320.5 to 666.8] | 349.2 [242.1 to 503.8] | 137.1 [82.0 to 229.1]
  HPV6 titers at Week 72 (n=55; 53; 53) | 112.8 [81.5 to 155.9] | 79.9 [52.1 to 122.6] | 43.0 [29.0 to 63.7]

6. Secondary Outcome: HPV11 Antibody Titers Among Those Seronegative for HPV11 at Baseline
Description: HPV antibody titers to type 11 were measured centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. The results below the lower limit of detection (LLD) were assigned the values of half the LLD (8 mMU/mL for HPV11). Geometric mean HPV11 titers with 95% CIs were calculated among the subset of participants who were seronegative for HPV11 (<16 mMU/mL) at baseline.
Time Frame: Weeks 28, 72
Population: All eligible participants who received at least one vaccine and were seronegative for HPV11 (HPV11-) at baseline (the number of participants analyzed) and had HPV11 titer available at the respective follow-up week. Strata A; B; C. Week 28: n=93; 70; 71. Week 72: n=83; 66; 69.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- Stratum A/Baseline HPV11-: Participants with screening CD4+ count >350 cells/mm^3 (Stratum A) who were seronegative for HPV11 at baseline.
- Stratum B/Baseline HPV11-: Participants with screening CD4+ count >200 to <=350 cells/mm^3 (Stratum B) who were seronegative for HPV11 at baseline.
- Stratum C/Baseline HPV11-: Participants with screening CD4+ count<=200 cells/mm^3 (Stratum C) who were seronegative for HPV11 at baseline.
Arm/Group | Stratum A/Baseline HPV11- | Stratum B/Baseline HPV11- | Stratum C/Baseline HPV11-
Number analyzed (Participants) | 99 | 72 | 74
mMU/mL
  HPV11 at Week 28 (n=93; 70; 71) | 476.5 [361.8 to 627.5] | 417.2 [286.8 to 606.8] | 205.1 [128.7 to 326.9]
  HPV11 at Week 72 (n=83; 66; 69) | 122.3 [90.1 to 166.0] | 85.1 [56.0 to 129.3] | 52.9 [35.0 to 79.9]

7. Secondary Outcome: HPV16 Antibody Titers Among Those Seronegative for HPV16 at Baseline
Description: HPV antibody titers to type 16 were measured centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. The results below the lower limit of detection (LLD) were assigned the values of half the LLD (11 mMU/mL for HPV16). Geometric mean HPV16 titers with 95% CIs were calculated among the subset of participants who were seronegative for HPV16 (<20 mMU/mL) at baseline.
Time Frame: Weeks 28, 72
Population: All eligible participants who received at least one vaccine and were seronegative for HPV16 (HPV16-) at baseline (the number of participants analyzed) and had HPV16 titer available at the respective follow-up week. Strata A; B; C. Week 28: n=73; 63; 64. Week 72: n=63; 59; 64.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- Stratum A/Baseline HPV16-: Participants with screening CD4+ count >350 cells/mm^3 (Stratum A) who were seronegative for HPV16 at baseline.
- Stratum B/Baseline HPV16-: Participants with screening CD4+ count >200 to <=350 cells/mm^3 (Stratum B) who were seronegative for HPV16 at baseline.
- Stratum C/Baseline HPV16-: Participants with screening CD4+ count<=200 cells/mm^3 (Stratum C) who were seronegative for HPV16 at baseline.
Arm/Group | Stratum A/Baseline HPV16- | Stratum B/Baseline HPV16- | Stratum C/Baseline HPV16-
Number analyzed (Participants) | 77 | 65 | 67
mMU/mL
  HPV16 at Week 28 (n=73; 63; 64) | 1199.9 [870.5 to 1654.1] | 1117.1 [746.2 to 1672.4] | 570.8 [327.7 to 994.3]
  HPV16 at Week 72 (n=63; 59; 64) | 248.9 [171.3 to 361.6] | 170.4 [106.8 to 271.8] | 98.3 [61.9 to 156.1]

8. Secondary Outcome: HPV18 Antibody Titers Among Those Seronegative for HPV18 at Baseline
Description: HPV antibody titers to type 18 were measured centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. The results below the lower limit of detection (LLD) were assigned the values of half the LLD (10 mMU/mL for HPV18). Geometric mean HPV18 titers with 95% CIs were calculated among the subset of participants who were seronegative for HPV18 (<24 mMU/mL) at baseline.
Time Frame: Weeks 28, 72
Population: All eligible participants who received at least one vaccine and were seronegative for HPV18 (HPV18-) at baseline (the number of participants analyzed) and had HPV18 titer available at the respective follow-up week. Strata A; B; C. Week 28: n=86; 80; 69. Week 72: n=75; 73; 69.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- Stratum A/Baseline HPV18-: Participants with screening CD4+ count >350 cells/mm^3 (Stratum A) who were seronegative for HPV18 at baseline.
- Stratum B/Baseline HPV18-: Participants with screening CD4+ count >200 to <=350 cells/mm^3 (Stratum B) who were seronegative for HPV18 at baseline.
- Stratum C/Baseline HPV18-: Participants with screening CD4+ count<=200 cells/mm^3 (Stratum C) who were seronegative for HPV18 at baseline.
Arm/Group | Stratum A/Baseline HPV18- | Stratum B/Baseline HPV18- | Stratum C/Baseline HPV18-
Number analyzed (Participants) | 92 | 83 | 73
mMU/mL
  HPV18 at Week 28 (n=86; 80; 69) | 175.0 [126.2 to 242.6] | 170.8 [114.5 to 254.7] | 93.6 [58.6 to 149.4]
  HPV18 at Week 72 (n=75; 73; 69) | 41.9 [29.5 to 59.0] | 40.6 [27.0 to 61.2] | 20.8 [14.5 to 30.0]

9. Secondary Outcome: Change in Log10 HPV6 Antibody Titers From Baseline Among Those Seropositive for HPV6 at Baseline
Description: Change in log10 HPV6 antibody titers was calculated as log10 HPV6 antibody titers at a later timepoint (Week 28, Week 72) minus log10 HPV6 antibody titers at baseline among those seropositive for HPV6 (>=20 mMU/mL) at baseline. HPV antibody titers to type 6 were measured centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. The results below the lower limit of detection (LLD) were assigned the values of half the LLD (7 mMU/mL, and after assay change in December 2012, 11 mMU/mL for HPV6).
Time Frame: Weeks 0, 28, 72
Population: All eligible participants who received at least one vaccine and were seropositive for HPV6 (HPV6+) at baseline (the number of participants analyzed) and had HPV6 titer available at the respective follow-up week. Strata A; B; C. Week 28: n=52; n=33; n=36. Week 72: n=43; 31; 35.
Measure: Median (Inter-Quartile Range); unit: Log10 mMU/mL
Groups:
- Stratum A/Baseline HPV6+: Participants with screening CD4+ count >350 cells/mm^3 (Stratum A) who were seropositive for HPV6 at baseline.
- Stratum B/Baseline HPV6+: Participants with screening CD4+ count >200 to <=350 cells/mm^3 (Stratum B) who were seropositive for HPV6 at baseline.
- Stratum C/Baseline HPV6+: Participants with screening CD4+ count<=200 cells/mm^3 (Stratum C) who were seropositive for HPV6 at baseline.
Arm/Group | Stratum A/Baseline HPV6+ | Stratum B/Baseline HPV6+ | Stratum C/Baseline HPV6+
Number analyzed (Participants) | 54 | 35 | 37
Log10 mMU/mL
  Change in HPV6 at Week 28 (n=52; 33; 36) | 1.12 [0.59 to 1.54] | 1.10 [0.61 to 1.52] | 0.97 [0.55 to 1.29]
  Change in HPV6 at Week 72 (n=43; 31; 35) | 0.73 [0.33 to 1.14] | 0.70 [0.41 to 1.00] | 0.44 [0.08 to 0.82]

10. Secondary Outcome: Change in Log10 HPV11 Antibody Titers From Baseline Among Those Seropositive for HPV11 at Baseline
Description: Change in log10 HPV11 antibody titers was calculated as log10 HPV11 antibody titers at a later timepoint (Week 28, Week 72) minus log10 HPV11 antibody titers at baseline among those seropositive for HPV11 (>=16 mMU/mL) at baseline. HPV antibody titers to type 11 were measured centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. The results below the lower limit of detection (LLD) were assigned the values of half the LLD (8 mMU/mL for HPV11).
Time Frame: Weeks 0, 28, 72
Population: All eligible participants who received at least one vaccine and were seropositive for HPV11 (HPV11+) at baseline (the number of participants analyzed) and had HPV11 titer available at the respective follow-up week. Strata A; B; C. Week 28: n=20; 21; 17. Week 72: n=17; 18; 19.
Measure: Median (Inter-Quartile Range); unit: Log10 mMU/mL
Groups:
- Stratum A/Baseline HPV11+: Participants with screening CD4+ count >350 cells/mm^3 (Stratum A) who were seropositive for HPV11 at baseline.
- Stratum B/Baseline HPV11+: Participants with screening CD4+ count >200 to <=350 cells/mm^3 (Stratum B) who were seropositive for HPV11 at baseline.
- Stratum C/Baseline HPV11+: Participants with screening CD4+ count<=200 cells/mm^3 (Stratum C) who were seropositive for HPV11 at baseline.
Arm/Group | Stratum A/Baseline HPV11+ | Stratum B/Baseline HPV11+ | Stratum C/Baseline HPV11+
Number analyzed (Participants) | 22 | 23 | 19
Log10 mMU/mL
  Change in HPV11 at Week 28 (n=20; 21; 17) | 1.32 [1.07 to 1.71] | 1.42 [0.86 to 1.59] | 0.60 [0.28 to 1.25]
  Change in HPV11 at Week 72 (n=17; 18; 19) | 0.93 [0.66 to 1.29] | 0.89 [0.64 to 1.14] | 0.43 [0.01 to 0.79]

11. Secondary Outcome: Change in Log10 HPV16 Antibody Titers From Baseline Among Those Seropositive for HPV16 at Baseline
Description: Change in log10 HPV16 antibody titers was calculated as log10 HPV16 antibody titers at a later timepoint (Week 28, Week 72) minus log10 HPV16 antibody titers at baseline among those seropositive for HPV16 (>=20 mMU/mL) at baseline. HPV antibody titers to type 16 were measured centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. The results below the lower limit of detection (LLD) were assigned the values of half the LLD (11 mMU/mL for HPV16).
Time Frame: Weeks 0, 28, 72
Population: All eligible participants who received at least one vaccine and were seropositive for HPV16 (HPV16+) at baseline (the number of participants analyzed) and had HPV16 titer available at the respective follow-up week. Strata A; B; C. Week 28: n=40; 28; 24. Week 72: n=37; 25; 24.
Measure: Median (Inter-Quartile Range); unit: Log10 mMU/mL
Groups:
- Stratum A/Baseline HPV16+: Participants with screening CD4+ count >350 cells/mm^3 (Stratum A) who were seropositive for HPV16 at baseline.
- Stratum B/Baseline HPV16+: Participants with screening CD4+ count >200 to <=350 cells/mm^3 (Stratum B) who were seropositive for HPV16 at baseline.
- Stratum C/Baseline HPV16+: Participants with screening CD4+ count<=200 cells/mm^3 (Stratum C) who were seropositive for HPV16 at baseline.
Arm/Group | Stratum A/Baseline HPV16+ | Stratum B/Baseline HPV16+ | Stratum C/Baseline HPV16+
Number analyzed (Participants) | 44 | 30 | 26
Log10 mMU/mL
  Change in HPV16 at Week 28 (n=40; 28; 24) | 1.65 [1.26 to 1.93] | 1.29 [0.84 to 1.86] | 1.06 [0.62 to 1.79]
  Change in HPV16 at Week 72 (n=37; 25; 24) | 1.28 [0.79 to 1.68] | 0.97 [0.56 to 1.59] | 0.53 [0.17 to 1.04]

12. Secondary Outcome: Change in Log10 HPV18 Antibody Titers From Baseline Among Those Seropositive for HPV18 at Baseline
Description: Change in log10 HPV18 antibody titers was calculated as log10 HPV18 antibody titers at a later timepoint (Week 28, Week 72) minus log10 HPV18 antibody titers at baseline among those seropositive for HPV18 (>=24 mMU/mL) at baseline. HPV antibody titers to type 18 were measured centrally using the competitive Luminex ImmunoAssay (HPV-4, cLIA) on stored serum. The results below the lower limit of detection (LLD) were assigned the values of half the LLD (10 mMU/mL for HPV18).
Time Frame: Weeks 0, 28, 72
Population: All eligible participants who received at least one vaccine and were seropositive for HPV18 at baseline (the number of participants analyzed) and had HPV18 titer available at the respective follow-up week. Strata A; B; C. Week 28: n=27; 11; 19. Week 72: n=25; 11; 19.
Measure: Median (Inter-Quartile Range); unit: Log10 mMU/mL
Groups:
- Stratum A/Baseline HPV18+: Participants with screening CD4+ count >350 cells/mm^3 (Stratum A) who were seropositive for HPV18 at baseline.
- Stratum B/Baseline HPV18+: Participants with screening CD4+ count >200 to <=350 cells/mm^3 (Stratum B) who were seropositive for HPV18 at baseline.
- Stratum C/Baseline HPV18+: Participants with screening CD4+ count<=200 cells/mm^3 (Stratum C) who were seropositive for HPV18 at baseline.
Arm/Group | Stratum A/Baseline HPV18+ | Stratum B/Baseline HPV18+ | Stratum C/Baseline HPV18+
Number analyzed (Participants) | 29 | 12 | 20
Log10 mMU/mL
  Change in HPV18 at Week 28 (n=27; 11; 19) | 1.02 [0.48 to 1.51] | 0.89 [0.50 to 1.53] | 0.85 [0.04 to 1.22]
  Change in HPV18 at Week 72 (n=25; 11; 19) | 0.57 [0.17 to 0.85] | 0.20 [-0.08 to 0.96] | 0.14 [0.02 to 0.61]

13. Secondary Outcome: Number of Participants With Signs and Symptoms of Grade 3 or Higher
Description: Number of participants who experienced a sign or symptom of Grade 3 or higher at any time after baseline while on study. Grading of signs and symptoms was according to Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004.
Time Frame: From baseline to up to Week 72
Population: All eligible participants who received at least one vaccine.
Measure: Number; unit: Participants
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 127 | 95 | 93
Participants | 20 | 20 | 16

14. Secondary Outcome: Number of Participants With Laboratory Abnormalities of Grade 3 or Higher
Description: Number of participants who experienced a laboratory abnormality of Grade 3 or higher at any time after baseline while on study. Grading of laboratory abnormalities was according to Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004.
Time Frame: From baseline to up to Week 72
Population: All eligible participants who received at least one vaccine.
Measure: Number; unit: Participants
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 127 | 95 | 93
Participants | 10 | 7 | 12

15. Secondary Outcome: Change in Log10 HIV Viral Load (VL) From Baseline
Description: A blood sample was drawn for local testing to determine the HIV VL. Change in log10 HIV VL was calculated as log10 HIV VL at a later time point (Weeks 4, 12, 28, 52 and 72) minus log10 HIV VL at baseline.
Time Frame: Weeks 0, 4, 12, 28, 52, and 72
Population: N=315 eligible participants who initiated intervention and had HIV VL available at Week 0 and the respective follow-up week. Strata A; B; C. Week 4: n=123; 89; 88. Week 12: n=118; 89; 90. Week 28: n=118; 91; 87. Week 52: n=109; 85; 82. Week 72: n=105; 81; 83.
Measure: Median (Inter-Quartile Range); unit: Log10 copies/mL
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 127 | 95 | 93
Log10 copies/mL
  Change in log10 HIV VL at Week 4 (n=123; 89; 88) | 0 [-0.18 to 0] | 0 [-0.06 to 0.11] | 0 [-0.15 to 0.01]
  Change in log10 HIV VL at Week 12 (n=118; 89; 90) | 0 [-0.27 to 0] | 0 [-0.21 to 0.09] | 0 [-0.45 to 0.23]
  Change in log10 HIV VL at Week 28 (n=118; 91; 87) | 0 [-0.43 to 0] | 0 [-0.63 to 0.12] | 0 [-0.46 to 0.17]
  Change in log10 HIV VL at Week 52 (n=109; 85; 82) | 0 [-0.53 to 0.08] | 0 [-1.11 to 0] | 0 [-1.28 to 0.44]
  Change in log10 HIV VL at Week 72 (n=105; 81; 83) | 0 [-0.59 to 0] | 0 [-1.03 to 0] | 0 [-1.93 to 0.15]

16. Secondary Outcome: Change in CD4 Cell Count From Baseline
Description: A blood sample was drawn for local testing to determine the CD4 cell count. Change in CD4 cell count was calculated as CD4 cell count at a later time point (Weeks 4, 8, 12, 24, 28, 52 and 72) minus CD4 cell count at baseline.
Time Frame: Weeks 0, 4, 8, 12, 24, 28, 52 and 72
Population: N=315 eligible participants who initiated intervention and had data available at Week 0 and the respective follow-up week. Strata A; B; C. Week 4: n=122; 92; 88. Week 8: n=119; 92; 90. Week 12: n=115; 87; 90. Week 24: n=117; 85; 88. Week 28: n=114; 89; 87. Week 52: n=108; 85; 87. Week 72: 105; 85; 88.
Measure: Median (Inter-Quartile Range); unit: Cells/mm^3
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 127 | 95 | 93
Cells/mm^3
  Change in CD4 count at Week 4 (n=122; 92; 88) | 31 [-52 to 94] | -3 [-45 to 29] | 5 [-13 to 29]
  Change in CD4 count at Week 8 (n=119; 92; 90) | 21 [-66 to 118] | -8 [-59 to 58] | 13 [-15 to 44]
  Change in CD4 count at Week 12 (n=115; 87; 90) | 5 [-99 to 104] | -3 [-42 to 63] | 13 [-19 to 47]
  Change in CD4 count at Week 24 (n=117; 85; 88) | 12 [-66 to 92] | 27 [-50 to 77] | 12 [-31 to 71]
  Change in CD4 count at Week 28 (n=114; 89; 87) | 35 [-60 to 113] | 37 [-49 to 104] | 17 [-25 to 72]
  Change in CD4 count at Week 52 (n=108; 85; 87) | 6 [-119 to 117] | 49 [-32 to 151] | 40 [-28 to 113]
  Change in CD4 count at Week 72 (n=105; 85; 88) | 31 [-91 to 93] | 65 [6 to 146] | 46 [-26 to 133]

ADVERSE EVENTS:
Time Frame: From baseline to up to Week 72
Description: The protocol required reporting of signs and symptoms and laboratory abnormalities of >=Grade 2 and all grades of fever. The DAIDS Adverse Event (AE) Grading Table, Version 1.0, December 2004 (Clarification, August 2009) was used for grading of AEs. Expedited adverse event reporting followed Version 2.0 of the DAIDS Expedited Adverse Event Manual.
Arm/Group | Stratum A | Stratum B | Stratum C
Serious Adverse Events (participants affected / at risk) | 6/127 | 2/95 | 6/93
Other Adverse Events (participants affected / at risk) | 96/127 | 71/95 | 82/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum A (N=127) | Stratum B (N=95) | Stratum C (N=93)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum A (N=127) | Stratum B (N=95) | Stratum C (N=93)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 11 | 8 | 12
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1 | 7
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 15
Leukoplakia oral (Gastrointestinal disorders) | 1 | 0 | 5
Nausea (Gastrointestinal disorders) | 14 | 6 | 15
Vomiting (Gastrointestinal disorders) | 13 | 4 | 16
Chest pain (General disorders) | 4 | 5 | 8
Chills (General disorders) | 5 | 2 | 5
Fatigue (General disorders) | 4 | 6 | 15
Injection site pain (General disorders) | 4 | 6 | 3
Oedema peripheral (General disorders) | 9 | 2 | 5
Pyrexia (General disorders) | 15 | 12 | 22
Bronchitis (Infections and infestations) | 10 | 5 | 4
Herpes simplex (Infections and infestations) | 5 | 3 | 5
Herpes zoster (Infections and infestations) | 0 | 7 | 2
Oral candidiasis (Infections and infestations) | 1 | 2 | 7
Upper respiratory tract infection (Infections and infestations) | 7 | 6 | 2
Urinary tract infection (Infections and infestations) | 9 | 6 | 7
Vaginitis bacterial (Infections and infestations) | 11 | 12 | 11
Vulvovaginal candidiasis (Infections and infestations) | 22 | 8 | 11
Vulvovaginitis trichomonal (Infections and infestations) | 5 | 5 | 1
Alanine aminotransferase increased (Investigations) | 2 | 7 | 6
Aspartate aminotransferase increased (Investigations) | 3 | 9 | 8
Blood bilirubin increased (Investigations) | 6 | 6 | 6
Blood creatinine increased (Investigations) | 4 | 1 | 10
Blood sodium decreased (Investigations) | 0 | 0 | 5
Haemoglobin decreased (Investigations) | 2 | 5 | 15
Neutrophil count decreased (Investigations) | 10 | 7 | 18
White blood cell count decreased (Investigations) | 0 | 2 | 14
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 8 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 0 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 10 | 11
Dizziness (Nervous system disorders) | 4 | 3 | 6
Headache (Nervous system disorders) | 17 | 11 | 13
Paraesthesia (Nervous system disorders) | 3 | 0 | 6
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 | 5 | 3
Anxiety (Psychiatric disorders) | 2 | 2 | 6
Depression (Psychiatric disorders) | 9 | 4 | 7
Insomnia (Psychiatric disorders) | 3 | 2 | 5
Dysuria (Renal and urinary disorders) | 7 | 1 | 5
Menorrhagia (Reproductive system and breast disorders) | 2 | 3 | 5
Vaginal discharge (Reproductive system and breast disorders) | 24 | 8 | 11
Vulvovaginal pruritus (Reproductive system and breast disorders) | 17 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 12 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Erythema (Skin and subcutaneous tissue disorders) | 2 | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 8 | 1 | 5
Hypertension (Vascular disorders) | 0 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.